CLINICAL TRIAL: NCT00700323
Title: Phase 2b Study of PS-Omega3 Conjugate Supplementation to ADHD Diagnosed Children
Brief Title: PS-Omega3 Supplementation to Attention Deficit Hyperactivity Disorder (ADHD) Children
Acronym: ADHD-3
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Enzymotec (Industry)
Responsible Party: Yoni Manor STUDY PROJECT MANAGER, Enzymotec Ltd.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TASMC-08-NV-263; 263-08-TLV
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Last update posted 2008-06-18 (Estimated); Status verified 2008-06

CONDITIONS: ADHD
Keywords: ADHD; ADHD diagnosed children
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients receiving active product
  Interventions: Dietary Supplement: PS-Omega3 conjugate supplementation
- 2 (Placebo Comparator): Patients receiving placebo
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: PS-Omega3 conjugate supplementation
  Arms: 1
Dietary Supplement: placebo
  Arms: 2

SUMMARY:
To assess the effect of phosphatidylserine-omega-3 consumption on the immune system parameters in children suffering from attention and concentration deficits.

ELIGIBILITY:
Inclusion Criteria:

1. Parental written informed consent.
2. Age: 13≥ years ≥8 (including).
3. Gender: both male and female.
4. TOVA computerized test score ≤-1.8 at baseline.
5. Language: Subjects, parents, and teachers must be able to read, write and speak Hebrew.
6. Normal weight and height according to Israeli standards.
7. 21 days without any treatment for ADHD symptoms, whether medication or food supplement.

Exclusion Criteria:

1. History or current diagnosis of any serious systemic (e.g., diabetes, hyper/hypothyroidism, etc.) or neurological condition (e.g., epilepsy, brain tumors, etc.)
2. Pervasive developmental disorder or Non-Verbal Learning Disability
3. Any evidence of psychotic disorders, suicidal risk, any current psychiatric co-morbidity that required psychiatric pharmacotherapy.
4. History of allergic reactions or sensitivity to marine products (seafood), soy or corn as well as any illness, which may jeopardize the participants health or limit their successful trial completion.
5. Having a sibling already included in the study.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nachum Vaisman, Prof', Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel